CLINICAL TRIAL: NCT00379756
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Study Evaluating the Efficacy, Safety, and Duration of Erection of Flexible-dose Vardenafil Administered for 12 Weeks Compared to Placebo in Subjects With Erectile Dysfunction and Dyslipidemia
Brief Title: A Study Evaluating Vardenafil Compared to Placebo in Subjects With Erectile Dysfunction (ED) and Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106718
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction, impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levitra (Active Comparator): 10mg x 4 weeks, with option to increase to 20mg aat that time if desired
  Interventions: Drug: LEVITRA (vardenafil)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LEVITRA (vardenafil) — active comparator
  Arms: Levitra
Drug: placebo — placebo comparator
  Arms: placebo

SUMMARY:
This is a study consisting of four periods (screening, run-in, treatment, follow-up). A four-week treatment-free, run-in period where the subject will make at least four attempts at intercourse on four separate days with at least 50% of the attempts must be unsuccessful. During run-in the subjects will be using a stopwatch to measure the time from erection perceived hard enough for penetration until withdrawal from the partner's vagina. Next there are 12 weeks of treatment with either placebo or LEVITRA. Each subject will be required to visit the clinic on 5 occasions over a period of 4 months.

ELIGIBILITY:
Inclusion criteria:

* Males with ED for more than six months, according to the NIH Consensus Statement (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance).
* Stable heterosexual relationship for more than 6 months.
* The subject must make at least four attempts at sexual intercourse (according to the question in the subject diary: Was sexual activity initiated with the intention of intercourse?) on four separate days during the untreated baseline period. At least 50% of attempts during this period must be unsuccessful, according to the following questions from the subject diary [at least one question should be answered "No"]: Were you able to achieve at least some erection (some enlargement of the penis)? Were you able to insert your penis into your partner's vagina? Did your erection last long enough for you to have successful intercourse?
* Diagnosis of dyslipidemia treated with a stable dose of a statin for 6 months at Visit 1.
* IIEF-EF domain score of 25 denoting mild to severe ED at Visit 2.
* Documented, dated, written Informed Consent.

Exclusion criteria:

* Premature ejaculator <2 minutes
* Any unstable medical, psychiatric, spinal cord injury, penile anatomical abnormalities, or substance abuse disorder that MD feels subject will not be able to complete the study.
* Low sexual desire.
* Prior prostatectomy surgery
* Severe chronic or acute liver disease, history of moderate or severe liver impairment
* Clinically significant chronic hematological disease
* Bleeding disorder or significant active peptic ulceration.
* Cardiovascular conditions that prevent sexual activity.
* History of heart attack, stroke, or life-threatening arrhythmia within the prior 6 months.
* hypotension or hypertension at rest.
* cancer within the past 5 years. Use of these medications: nitrates or nitric oxide donors, anti-androgens, oral or injectable androgens, received any investigational drug (including placebo) within 30 days of screening (Visit 1).
* Use of any treatment for ED within 7 days of screening including oral medications, vacuum devices, constrictive devices, injections or urethral suppositories.
* Subjects who are taking the following potent inhibitors of cytochrome P-450 3A4.
* Abnormal Laboratory Values:

  1. serum total testosterone level >25% below the lower limit of normal
  2. serum creatinine >3.0 mg/dl.
  3. AST and/or ALT >3x the upper limit of normal.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 395 (Actual)
Dates: Start 2006-05-22 (Actual); Primary Completion 2007-05-17 (Actual); Study Completion 2007-05-17 (Actual)

PRIMARY OUTCOMES:
Erectile function (EF) domain score of the International Index of Erectile Function (IIEF) | Up to Week 12
  The IIEF questionnaire is a validated 15-item instrument that assesses the participant's erectile function over the previous 4 weeks. The IIEF includes 5 domains affecting male sexual function: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Responses to the IIEF were re-coded using a standard coding method, where more positive responses received a higher score. The EF domain score was calculated as the sum of the re-coded scores from questions 1-5 and 15, using last observation carried forward (LOCF). Scores range from 1 (lowest) to 30 (highest). If two or more items in the EF domain were missing, the EF domain score was considered to be missing.
Mean success rate of insertion based on attempts | Up to Week 12
  Success rate of insertion was derived from the Sexual Encounter Profile (SEP) Question 2 (SEP-2) of the participant's diary that asked 'Were you able to insert your penis into your partner's vagina?'. Responses were either Yes or No. Patients were instructed to complete diary questions as soon as possible after each sexual attempt, but no later than 24 hours after the attempt. The per-participant overall success rate for insertion was calculated by dividing the number of successful attempts (SEP-2=yes) over 12 weeks by the total number of valid attempts recorded over 12 weeks. If the participant was not able to make any valid attempts in 12 weeks, the participant was non-evaluable. Per-participant success rates were then averaged at the group level to obtain the mean success rate from Weeks 0-12.
Mean success rates of maintenance based on attempts | Up to Week 12
  Success rate of maintenance was derived from the SEP Question 3 (SEP-3) of the participant's diary that asked 'Did your erection last long enough for you to have successful intercourse?'. Responses were either Yes or No. Participants were instructed to complete diary questions as soon as possible after each sexual attempt, but no later than 24 hours after the attempt. The per-participant overall success rate for maintenance was calculated by dividing the number of successful attempts (SEP-3=yes) over 12 weeks by the total number of valid attempts recorded over 12 weeks. If the participant was not able to make any valid attempts in 12 weeks, the participant was non-evaluable. Per-participant success rates were then averaged at the group level to obtain the mean success rate from Weeks 0-12.

SECONDARY OUTCOMES:
Mean duration of erection leading to completion of successful intercourse as measured by Sexual Encounter Profile Question 3 [SEP-3] | Up to Week 12
  Duration of erection leading to completion of successful intercourse was derived from data recorded in the participant's diary. For each diary entry, the time from erection perceived hard enough for penetration until withdrawal from partner's vagina was measured by stopwatch and recorded in the participant's diary. For diary entries where SEP-3=yes, this recorded duration was used in calculations of a per-participant median duration. For diary entries where SEP-3=no, a duration of 0 was used to calculate the per-participant median. The per-participant median values averaged at the group level to obtain the mean duration of erection leading to completion of successful intercourse as measured by SEP-3.
Change from Baseline in scores for questions on the IIEF questionnaire and scores of the other non-EF domains of the IIEF | Up to Week 12
  Non-EF domains of the IIEF (Intercourse Satisfaction, Orgasmic Function, Sexual Desire, Overall Satisfaction) and IIEF questions (Erection during sexual activity?, Hard enough for penetration?, Able to penetrate partner?, Maintain your erection?, Maintain to completion?, Times attempted intercourse, Satisfactory for you?, Enjoyed sexual intercourse?, How often did you ejaculate?, How often feeling of orgasm?, How often felt sexual desire?, Rate level of sexual desire?, How satisfied with sex life?, Satisfied with sexual relationship? and Confidence to get, keep erection?) scores were assessed at Week 4, Week 8 and Week 12. The Baseline was the value at Week 0. Change from Baseline was the post-Baseline value minus Baseline value.
Number of participants with normal erectile function having EF domain scores of 26 and above | Up to Week 12
  The EF domain score was calculated by summing recoded responses to Questions 1-5 and 15, for each participant. It ranged from 1 to 30. EF domain scores were dichotomized as either normal (26 and above) or below normal (below 26) using LOCF, to calculate number of participants returning to normal erectile function. For the EF domain score the total was considered to be missing if 2 or more answers in the domain were missing.
Change from Baseline in participant's diary results | Up to Week 12
  Electronic diaries were provided to participants. Participants were supposed to complete the diary questions as soon as possible after each sexual attempt but no later than 24 hours after the attempts. The diary questions (Ability to achieve at least some erection, Ability to insert penis into partner's vagina, Long enough erection having successful intercourse, Satisfied with the hardness of erection, Satisfied with this sexual experience, Ability to ejaculate) response rates were presented for Weeks 0-12. The Baseline was the value at Week 0. Change from Baseline was the post-Baseline value minus Baseline value.
Mean duration of erection regardless of SEP-3 Response | Up to Week 12
  Duration of erection was time from erection perceived hard enough for penetration (start stopwatch) until withdrawal from the partner's vagina (stop stopwatch) regardless of completion of successful intercourse. The data was presented for overall period from Week 0 to Week 12.
Change from Baseline in duration of erection leading to completion of successful intercourse. | Up to Week 12
  Duration of erection was time from erection perceived hard enough for penetration (start stopwatch) until withdrawal from the partner's vagina (stop stopwatch) leading to completion of successful intercourse. The data was presented for overall period from Week 0 to Week 12. The Baseline was the value at Week 0. Change from Baseline was the post-Baseline value minus Baseline value.
Number of participants with response 'Yes' for Global Assessment Question | Up to Week 12
  The participants were asked to complete the self-administered Global Assessment Question. The question asked was 'has the treatment you have been taking over the past 4 weeks improved your erections'. The response was either Yes or No depending on comparison to participant's erections before their participation in this study. For the scale missing values remained missing.
Mean score for Keep It Simple (KIS) scale | Up to Week 12
  The KIS scale was a self-reported visual analog scale (VAS) from 0 to 10 designed to assess erections as 'how do you grade your erections over the last 4 weeks?'. For the scale missing values remained as missing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- United States (64):
  - GSK Investigational Site, Fairhope, Alabama
  - GSK Investigational Site, Homewood, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Orangevale, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Pinecrest, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Dawsonville, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Swansea, Maine
  - GSK Investigational Site, Taunton, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Lawrenceville, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, West Seneca, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Shippensburg, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Menomonee Falls, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin